CLINICAL TRIAL: NCT06014411
Title: Early Versus Delayed Bathing of Orthopaedic Surgical Wounds: a Prospective Randomized Controlled Study
Brief Title: Early Versus Delayed Bathing of Orthopaedic Surgical Wounds
Acronym: EVDB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: New York Presbyterian Hospital (Other)
Responsible Party: Principal Investigator, William Ricci, Chief Orthopaedic Trauma Service, Hospital for Special Surgery, New York
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2023-1723; 21-04023565 (Other: Weill Cornell Medicine IRB #)
Record Dates: First submitted 2023-08-21; First posted 2023-08-28 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Surgical Wound; Post Operative Wound Infection
MeSH Terms: conditions — Surgical Wound; Surgical Wound Infection

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Delayed Bathing (Active Comparator): Delayed bathing-- patients will be told to begin showering after wound exam and suture removal (10-20 day postoperative).
  Interventions: Other: Time to bathing (delayed)
- Early Bathing (Active Comparator): Early bathing--Patients will be told to remove dressings and begin showering with body soap on postoperative day 3.
  Interventions: Other: Time to bathing (early)

INTERVENTIONS:
Other: Time to bathing (delayed) — Delayed bathing-- patients will be told to begin showering after wound exam and suture removal (10-20 day postoperative).
  Arms: Delayed Bathing
Other: Time to bathing (early) — Early bathing--Patients will be told to remove dressings and begin showering with body soap on postoperative day 3.
  Arms: Early Bathing

SUMMARY:
This is a single center randomized control trial assessing the effect of early versus delayed bathing on orthopaedic surgical wounds in patients undergoing surgical treatment of fractures. Patients will be recruited by screening all patients undergoing surgical treatment for fractures at our institution. Patients who provide written consent will be randomized to one of two treatment arms after confirming eligibility criteria. Group A will be advised to begin early normal bathing (non-submerged showering) with uncovered surgical wounds. Group B will be advised to follow traditional delayed bathing with covered wounds.

Those who do not wish to participate in the randomized trial will be invited to participate observationally (no randomization) and have the same prospective follow-up.

DETAILED DESCRIPTION:
The study is a single center, non-inferiority, parallel group, randomized control trial assessing the effect of early versus delayed bathing on orthopaedic surgical wounds in patients undergoing surgical treatment of fractures. Patients will be recruited by screening all patients undergoing surgical treatment for fractures at our institution. Patients who provide written consent will be randomized to one of two treatment arms after confirming eligibility criteria. Group A will be advised to begin early normal bathing (non-submerged showering) with uncovered surgical wounds. Group B will be advised to follow traditional delayed bathing with covered wounds.

Patients will have follow-up with data collection at two, six and 12 weeks post-operatively. The primary outcome measure will be patient satisfaction as measured by a Likert Scale. The Likert Scale as utilized will be a patient reported outcome measure consisting of one question allowing the subject to express their attitude towards a particular subject: "How satisfied are you with your surgical treatment" with possible answers consisting of: "very satisfied", "somewhat satisfied", "neutral", "somewhat unsatisfied", and "very unsatisfied". The secondary outcome measures will be development of an infection (subcategorized as either superficial or deep) and development of peri-incisional inflammation (eg. adhesive rash).

Primary Objective: The primary objective of the study is to compare patient satisfaction as measured using a Likert Scale associated with early and delayed surgical site bathing.

Secondary Objectives: The secondary objective is to compare the infection rate of orthopaedic surgical wounds between early and delayed bathing.

Those who do not wish to participate in the randomized trial will be invited to participate observationally (no randomization) and have the same prospective follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patient who are not pregnant
* Isolated acute fractures of the upper or lower extremities (humerus, radius, ulna, femur, tibia, or fibula)
* Diagnosis of a fracture meeting indication for operative intervention
* Any fracture not requiring a splint for post-operative management
* Non-complicated wounds (non-traumatic wounds, closed injuries, fractures not requiring external fixation, and acute fracture surgery)

Exclusion Criteria:

* Fractures associated with presumed infection
* Patients with multiple fractures
* Fractures in patients with underlying associated immune compromise
* Fractures in patients with underlying peripheral vascular disease
* Use of VAC
* Surgery performed through previous surgical wound
* Patient homeless
* Fractures in patients with underlying diabetes mellitus
* Complicated wounds (traumatic wounds, need for post-op wound care, open injuries, need for external fixation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction associated with early and delayed surgical site bathing | Weeks 2, 6 and 12 post surgery
  The primary endpoint of the study will be a statistically significant difference in patient satisfaction as measured using a Likert Scale between the two groups. Scale will be on scale 0-10. A score of 10 will be "Very Satisfied" and a score of 0 will be "Very Dissatisfied."

SECONDARY OUTCOMES:
Infection rate of orthopaedic surgical wounds between early and delayed bathing | Weeks 12 post surgery
  The secondary endpoint in this study will be a statistically significant or clinically important difference in infection rate of orthopaedic surgical wounds between the early and delayed bathing groups

CONTACTS AND LOCATIONS:
Overall Officials: William M Ricci, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- NewYork-Presbyterian/Weill Cornell Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided